CLINICAL TRIAL: NCT05085067
Title: The Efficacy of Auto-crosslinked Hyaluronic Acid Gel in the Prevention of Adhesion Reformation After Hysteroscopic Resection of Retained Products of Conception:a Randomized Controlled Trial
Brief Title: The Efficacy of Auto-cross Linked Hyaluronic Acid Gel in the Prevention of Adhesion Reformation After Hysteroscopic Resection of Retained Products of Conception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Yang Xue, principal investigator, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FXHV1.0-2020-11-15
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Retained Products of Conception
Keywords: Retained Products of Conception; Hysteroscopy; Intrauterine adhesion; Auto-crossed-linked hyaluronic acid gel
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: no auto-cross linked hyaluronic acid gel (No Intervention): no auto-cross linked hyaluronic acid gel into intrauterine cavity after hysteroscopic treatment because of retained products of conception
- Group B: infusing auto-cross linked hyaluronic acid gel (Experimental): infusing auto-cross linked hyaluronic acid gel into intrauterine cavity after hysteroscopic treatment because of retained products of conception
  Interventions: Other: auto-crossed-linked hyaluronic acid gel

INTERVENTIONS:
Other: auto-crossed-linked hyaluronic acid gel — infusing auto-cross linked hyaluronic acid gel into intrauterine cavity after hysteroscopic treatment because of retained products of conception
  Arms: Group B: infusing auto-cross linked hyaluronic acid gel

SUMMARY:
Retained product of conception (RPOC) is defined by abnormal trophoblastic persistence or retained placenta inside the uterus cavity after a pregnancy independently of the outcome. Untreated RPOC can compromise future fertility. RPOC are generally treated surgically, either by repeated evacuation or by hysteroscopy, which exposes the uterus to additional potential trauma.The combination of trauma to the gravid uterine cavity, hypoestrogenic state at the time of the operation or immediately afterward and local infection is considered to be the pathogenic mechanism of intrauterine adhesions (IUA) , manifested clinically by menstrual abnormalities, infertility and recurrent pregnancy loss.To investigate the efficacy of auto-cross linked hyaluronic acid gel in the prevention of adhesion reformation after hysteroscopic resection of retained products of conception.

After the completion of hysteroscopic resection of retained products of conception, patients will be randomized to one of the two groups by computer-generated numbers: [1] infusing auto-cross linked hyaluronic acid gel into intrauterine cavity in the experimental group; [2] no auto-cross linked hyaluronic acid gel into intrauterine cavity in the control group. Second and third look outpatient hysteroscopy will be performed 4 and 8 weeks after the initial surgery. The patients will be followed up about menstrual pattern at 3 months after the surgery.The patients will be followed up about pregancy outcome at 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of retained products of conception
* Written consent obtained

Exclusion Criteria:

* Patients with severe complications of medicine and surgery
* Acute or chronic genital tract inflammation
* No understanding or approving the randomized controlled trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Adhesion reformation rate at third-look hysteroscopy | A third-look hysteroscopy will be carried out 8 weeks after the initial operation.Findings are graded according to the American Fertility Society classification.
Adhesion score at third-look hysteroscopy | A third-look hysteroscopy will be carried out 8 weeks after the initial operation.Findings are graded according to the American Fertility Society classification.
Concentration of the menstrual pattern | at 3 months after the initial surgery
Pregnancy rate | at 12-month after the initial surgery

SECONDARY OUTCOMES:
Rate of complications | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- FuxingHospital，Captital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided